CLINICAL TRIAL: NCT00077961
Title: Phase I/II Study of Rituximab Plus CAMPATH in Patients With Previously Treated Relapsed or Refractory Low-Grade Follicular, CD20-positive, B-cell Non-Hodgkin's Lymphoma
Brief Title: Rituximab Plus CAMPATH in Patients With Relapsed/Refractory Low-Grade or Follicular, CD20-positive, B-cell NHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM.NHL233
Record Dates: First submitted 2004-02-13; First posted 2004-02-18 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; NHL; CAMPATH; alemtuzumab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Alemtuzumab

INTERVENTIONS:
Drug: CAMPATH (alemtuzumab)

SUMMARY:
The purpose of this study is to determine the optimal dose of subcutaneous CAMPATH when used in combination with rituximab for patients with relapsing or refractory, low-grade or follicular, CD-20-positive, B-Cell non-Hodgkin's Lymphoma. Safety will be the primary objective of phase I, while the primary objective of phase II will be to determine overall response.

DETAILED DESCRIPTION:
This study is being conducted in 2 parts. Phase I will involve dose escalation of subcutaneous CAMPATH (SQ) given 3 times per week in combination with weekly doses of rituximab (375mg/m2) for a maximum of 8 weeks in order to determine the maximum tolerated dose (MTD). In Phase II patients will be treated with SQ CAMPATH at the MTD plus weekly rituximab (375mg/m2)for a maximum of 8 weeks with primary objective of defining Overall Response (OR) to this combination.

ELIGIBILITY:
Inclusion Criteria:

* For the Phase I portion of the study, patients must have pathologically confirmed diagnosis of low-grade or follicular, CD20-positive, B-cell, non-Hodgkin's lymphoma that has relapsed or is refractory. For the Phase II portion of the study, patients must have a pathologically confirmed diagnosis of low-grade or follicular, CD20-positive, B-cell, non-Hodgkin's lymphoma (Follicular, predominantly small cleaved or follicular, mixed small cleaved and large cell, International Working Formulation classification B or C or REAL classification follicular center grade 1,2) that has relapsed or is refractory.
* Previously treated with at least one anti-cancer regimen for NHL
* Measurable disease (lesions that can be accurately measured in 2 dimensions by CT scan with a greatest transverse diameter of >/= to 2cm or palpable lesions with both diameters of 2cm or more)
* Life expectancy of at least 12 weeks
* WHO performance status or 0 or 1
* Adequate marrow and organ function (as defined in the protocol)
* Completed major surgery, radiotherapy, chemotherapy, immunotherapy or biotherapy/targeted therapies at least 4 weeks prior to study entry (6 weeks if treated with a nitrosourea or mitomycin). Patients must have recovered from all prior treatment toxicity to Grade 1 or less, exclusive of alopecia.

Exclusion Criteria:

* Prior combination therapy with rituximab and CAMPATH; prior therapy with either agent alone is permitted
* A history of a T-cell lymphoma
* Known AIDS-related HIV-positive lymphoma
* For the Phase II portion of the study (once MTD has been determined), bulky disease, ie, any single mass >10cm or circulating malignant cells of 25,000/uL or more
* Prior autologous bone marrow or stem cell transplant within 6 months of study entry
* Prior allogeneic bone marrow transplant or organ transplant
* Prior radiotherapy to the only site of measurable disease
* Medical condition requiring chronic use of oral, high-dose corticosteroids
* Use of investigational agents within 30 days of study enrollment
* Past history of anaphylaxis following exposure to humanized monoclonal antibodies
* Known, active, infection, including HIV positive
* Diagnosis of another malignancy within the previous five (5) years, unless the probability of recurrence of the prior malignancy is < 5%. Patients with curatively treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, cervical intraepithelial neoplasia (CIN), and patients with a history of malignant tumor in the past that have been disease-free for at least 5 years
* Active central nervous system (CNS) involvement with lymphoma
* Pregnant or nursing women
* Any significant concurrent disease or illness that would, in the opinion of the investigator, compromise patient safety or compliance, or interfere with the interpretation of study results
* Active hepatitis or a history of prior viral hepatitis B or C, or positive hepatitis B serologies without prior immunization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49
Dates: Start 2003-12; Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (10):
- United States (10):
  - Colorado Springs, Colorado
  - Ocala, Florida
  - Park Ridge, Illinois
  - Lafayette, Louisiana
  - New Orleans, Louisiana
  - Columbia, Missouri
  - Manhasset, New York
  - Cary, North Carolina
  - Canton, Ohio
  - Greenville, South Carolina